CLINICAL TRIAL: NCT06880237
Title: Sing Out Loud: a Choral Singing Program for Persons Living with Dementia
Acronym: SOL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Collaborators: Esplanade (Unknown); APEX Harmony Lodge (Unknown)
Responsible Party: Principal Investigator, Kathleen Rose Agres, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NUS-IRB-2023-164
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Dementia; Nursing Homes Residents
Keywords: Dementia; Nursing Home Residents; Singing; Biomarkers; NPI-Q
MeSH Terms: conditions — Dementia | interventions — Singing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Singing group (Experimental): The intervention for the Singing group will be the 8-week SOL programme.
  Interventions: Other: Singing
- Waitlist Control group (No Intervention): The Waitlist Control group will not receive any intervention during the course of the study but will receive the SOL programme in its next iteration.

INTERVENTIONS:
Other: Singing — The programme consists of nin 75-min-long singing sessions spread across 8 weeks (8 sessions are practice sessions and 1 session is a full dress rehearsal), and a final performance. The final rehearsal session and showcase performance will be held at a concert venue, while the 8 practice sessions will be conducted at the nursing home.
  Each session will kick off with a "Hello song", followed by warm-up activities and vocal exercises. Participants will then sing different songs to explore and rehearse as a group, before concluding with a "Goodbye song". All sessions throughout the programme are similarly structured to provide consistency for participants.
  Arms: Singing group

SUMMARY:
We intend to investigate whether a singing programme for nursing home residents living with dementia can reduce the mental and physiological effects of dementia. The main questions it aims to answer are:

1. Does participating in the Sing Out Loud (SOL) singing intervention lead to an improvement in the physiological well-being (increase in oxytocin and reduction in cortisol levels) of persons living with dementia (PWDs) in nursing homes?
2. Will participation in the SOL singing intervention result in an improvement in PWDs' overall mood, temperament, and mental health (indicated by symptoms such as apathy, aggression, and depression).

Researchers will compare the singing group to the control group to see if they exhibit reduced levels of apathy, aggression, and depression, and whether their levels of oxytocin and cortisol (collected via salivary biomarkers) have increased and decreased, respectively.

Researchers will compare the SOL singing intervention with a waitlist control group to see if the SOL singing intervention increases the feelings of social connection, reduces stress, or improves the symptoms of dementia in nursing home residents.

Participants will be randomly assigned to a singing intervention or waitlist control group. The intervention involves an 8-week long singing programme with one practice session a week, culminating in an additional full dress rehearsal and private showcase performance for their family members at a concert venue.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Aged 59 to 90 years old
* Diagnosed with dementia
* Living in the nursing home
* Interested in participating in the SOL programme
* Able to provide saliva samples

Exclusion Criteria for Patients:

* Unable to provide saliva samples

Inclusion Criteria for Psychologists:

* Aged 21 to 65 years old
* Is the psychologist of a patient who is participating in the SOL programme
* Is able to speak English

Exclusion Criteria for the Psychologists:

* Unable to complete the NPI-Q questionnaire for their patient who is participating in the SOL programme
* Decline audio recording during the focus group discussion

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-03-12 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in Oxytocin and Cortisol levels at 8 weeks | From the beginning of the intervention (session 1) on week 1, to the final practice session (session 8) on week 8
  Oxytocin and Cortisol levels will be collected via saliva samples. Increases in level of Oxytocin is indicative of increased feelings of social connection, while increased level of Cortisol is indicative of higher levels of stress
Change from baseline in the severity and distress of neuropsychiatric symptoms at 8 weeks | From 2 weeks before session 1, up to the final practice session (session 8)
  Neuropsychiatric symptoms will be collected via the Neuropsychiatric Inventory Questionnaire (NPI-Q), which measures delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability, motor disturbance, nightime behaviours, and appetite. Higher scores indicate increased levels of severity or distress related to the symptom in question.

SECONDARY OUTCOMES:
Qualitative feedback | Within two weeks after the programme has ended
  This will be collected via a focus group discussion with the nursing home's clinical staff (psychosocial team) to collect qualitative data on any observed changes in participants' mood, behaviour, temperament, or relationships between participants and staff. Additionally, they will also be asked about process factors (challenges in implementation, structure and delivery of the programme), satisfaction,

CONTACTS AND LOCATIONS:
Locations (1):
- APEX Harmony Lodge, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No